CLINICAL TRIAL: NCT02332759
Title: A PILOT STUDY TO EVALUATE THE PRELIMINARY SAFETY AND FEASIBILITY OF THE MATERNA MEDICAL DEVICE FOR THE PREVENTION OF PERINEAL LACERATIONS AND OCCULT DISRUPTION OF THE PELVIC FLOOR AND ASSOCIATED SEQUELA DURING VAGINAL DELIVERY.
Brief Title: A Pilot Study To Evaluate The Preliminary Safety And Feasibility Of The Materna Medical Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Materna Medical (Industry)
Responsible Party: Principal Investigator, Francisco Orejuela, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H- 31936
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Tear, Pelvic Organ, Obstetric Trauma
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Materna Device (Experimental): The device will be inserted vaginally for one hour during active phase of labor to dilate the vaginal canal.
  Interventions: Device: Materna Medical

INTERVENTIONS:
Device: Materna Medical

SUMMARY:
The Materna device aims to prevent pelvic tissue damage by preventing overstretching of pelvic floor muscle fibers during delivery. The device is a single use, disposable, mechanical dilator that penetrates the first 4 cm or ½ of the vaginal canal and gradually expands the vagina from a resting diameter of 2-3 cm to the fully expanded size of a delivering fetus, roughly 8-10 cm. The Materna device will be used during the first stage of labor, for roughly 1-2 hours, in a hospital Labor and Delivery unit, under the supervision of trained clinical labor and delivery providers

DETAILED DESCRIPTION:
Over 80% of women who deliver vaginally will sustain a vaginal tear, and roughly half of all women will suffer from permanent pelvic muscle damage that may lead to pelvic disorders later in life.(1-8) The consequences of vaginal tearing are acute and chronic pain, longer recovery times, sexual dysfunction and permanent disfigurement.(1-4) Additionally, women often say that the prospect of tearing is one the things they fear most regarding childbirth. Tearing during childbirth is well documented as occurring during most deliveries, however there is additional damage now being discovered that occurs internally to the pelvic muscles.

It has long been thought that childbirth is the leading factor contributing to the development of pelvic floor disorders such as pelvic organ prolapse, urinary and fecal incontinence. (6,9,10) In the last 10 years, new imaging studies have shown that approximately 20-30% of women will have their pelvic muscles permanently separated from the pelvic bone during vaginal delivery.(5-11) In an additional 20-30% of cases, the muscles may remain attached to the pelvic bone but have been stretched to the point of becoming functionally compromised

One of the most promising ideas to prevent this damage is to slowly prepare the pelvic muscles, during labor while the cervix is dilating, in order to maximize their stretch.

The previous data and preliminary findings of Materna suggest the following overall working hypotheses:

1. Vaginal lacerations and pelvic floor muscle damage lead to increased incidence of pelvic floor disorders and other negative sequelae.
2. Vaginal lacerations and pelvic floor muscle damage are caused by over straining of pelvic muscles and vaginal tissues without maximizing the tissue strain using appropriate viscoelastic relaxation during the second phase of labor.
3. The incidence and severity of vaginal lacerations and pelvic floor muscle damage can be reduced by inducing a more gradual strain of the vaginal tissues using a device-based approach

Currently there are no devices available in the U.S. to protect the pelvic muscles from damage during childbirth. The Materna device takes advantage of well-proven biomechanical data in the fields of sports medicine and orthopedics showing that tissue is viscoelastic, meaning that the more slowly it is stretched the easier it is to stretch. Materna aims to take advantage of this biomechanical phenomena as well as the length of the first phase of labor to reduce the tension in the tissue, slowly maximizing the stretch of the tissue in order to prepare it for a delivery with less injury. There is also evidence showing that reducing the tension in the pelvic muscles could lead to a shorter delivery time, resulting in a less stressful and healthier delivery for the baby

ELIGIBILITY:
Inclusion Criteria:

* Primiparas, or previous pregnancy terminated before 24 weeks gestation
* Single fetus birth
* Subject is able to understand the risks and potential benefits of participating in the study and is willing to provide written informed consent
* Subject is willing and able to comply with specified follow-up evaluations
* Planned to have epidural during birthing process

Exclusion Criteria:

* Previous delivery, or previous pregnancy beyond 24 weeks gestation
* Less than 36 weeks gestation
* Neurological diseases e.g. Multiple Sclerosis that may result in unrelated pelvic disorders
* Muscular or skin disorder that effects elasticity of tissue such as scleroderma or lupus
* Local or systemic infection e.g. HIV, herpes
* Diabetes
* Clinically estimated fetal weight > 4,500 grams
* Any prior surgical procedures to the vaginal anatomy which could lead to pelvic dysfunction, pelvic fractures, or pelvic soft tissue injuries. Evaluated during baseline screening
* High likelihood of less than 1 hour of potential device dilation time after the woman arrives at the center and receives epidural
* A cervical dilation of greater than or equal to 6 cm
* BMI > 32.5 prior to becoming pregnant

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
No adverse events related to device | 12-20 week postpartum follow up

SECONDARY OUTCOMES:
Reduction in perineal lacerations and pelvic floor trauma | 12-20 week postpartum follow up

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Ramin, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital Pavilion For Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No